CLINICAL TRIAL: NCT02884895
Title: Establishing a Definitive Airway: A Comparison of Direct Laryngoscopy With Blind Intubation Via Intubating Laryngeal Tube Suction Disposable
Brief Title: A Comparison of Direct Laryngoscopy With Blind Intubation Via Intubating Laryngeal Tube Suction Disposable
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-007
Record Dates: First submitted 2016-08-16; First posted 2016-08-31 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-08

CONDITIONS: Adverse Anesthesia Outcome
Keywords: Intubating Laryngeal Tube Suction; Blind intubation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intubating laryngeal Tube Suction (Experimental): Intubating laryngeal Tube Suction
  Interventions: Device: Intubating Laryngeal Tube Suction
- Direct Laryngoscopy (Active Comparator): Direct Laryngoscopy
  Interventions: Device: Direct Laryngoscopy

INTERVENTIONS:
Device: Intubating Laryngeal Tube Suction — Intubating Laryngeal Tube Suction Disposable
  Arms: Intubating laryngeal Tube Suction
Device: Direct Laryngoscopy — Direct Laryngoscopy
  Arms: Direct Laryngoscopy

SUMMARY:
Tracheal intubation is an important part of treatment for a trauma casualty. Tracheal intubation is usually achieved by a direct laryngoscope.It is an effective method but requires experience and skill demanding a long learning time.The use of the Laryngeal Tube Suction for fast control of the airway is known for many years. The Intubating Laryngeal Tube Suction is a new version of the Laryngeal Tube. The aim of this study is to examine the effectiveness of the the Intubating Laryngeal Tube Suction to achieve a definitive airway by unskilled practitioners in anesthetized patients with the head in neutral position (trauma model).

DETAILED DESCRIPTION:
Control the airways and respiration are an important part of treatment for a trauma casualty. Tracheal intubation an action that allows the insertion of a tube through the vocal cords and fixation by the balloon inflation is a definitive airway.

Tracheal intubation is usually achieved by a direct laryngoscope. This method is taught both in the training of doctors and paramedics training. Although it is an effective method requires experience and skill demanding a long learning time The use of the Laryngeal Tube Suction for fast control of the airway is known for many years. The Laryngeal Tube Suction and others similar devices are known as Supraglottic Airway Devices and are inserted blind in the oropharynx and allow a fast oxygenation and ventilation of the patients.

The new generation of these devices allows perform blind intubation directly through a special channel. One of these devices is the Intubating Laryngeal Tube Suction

The aim of this study is to examine the effectiveness of the Intubating Laryngeal Tube Suction to achieve a definitive airway by unskilled practitioners in anesthetized patients with the head in neutral position (trauma model).

The hypothesis is that definitive airway obtaining with Intubating Laryngeal Tube Suction will be more success and faster compared to the standard way of direct laryngoscope. If the hypothesis is proven, this research will be very important implications for the management of the airway describing pre-hospital and in particular military scenarios.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology class I and II

Exclusion Criteria:

* Difficult airways
* Cervical pathology
* Full stomach

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Blind tracheal intubation time measure in seconds | 30 seconds

SECONDARY OUTCOMES:
Easy of insertion measure in numerical scale | 30 seconds
  Easy of insertion measure 1 to 5 Numerical scale

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Gaitini, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes